CLINICAL TRIAL: NCT01764880
Title: Phase I Dose Finding Study Assessing Safety and Tolerability of SST0001 in Advanced Multiple Myeloma.
Brief Title: SST0001 (Roneparstat) in Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sigma Tau Research Switzerland SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SST0001-STRCH-CR-11-002
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
Keywords: Heparanase inhibitor; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — SST 0001; roneparstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SST0001 (Roneparstat) (Experimental): SST0001 once daily for 5 or 10 days in a cycle of 28 days. Starting dose 25 mg, to be escalated in subsequent cohorts.
  Duration of treatment depending on toxicities observed or until documentation of disease progression or other discontinuation criteria are met.
  Interventions: Drug: SST0001 (Roneparstat)

INTERVENTIONS:
Drug: SST0001 (Roneparstat) — SST0001 once daily for 5 or 10 days in a cycle of 28 days.

SUMMARY:
Heparanase cleaves heparan sulfate (HS) chains, a natural substrate for heparanase, and participates in degradation and remodelling of the extra-cellular matrix (ECM) facilitating, among other activities, cell invasion associated with cancer metastasis, angiogenesis, and inflammation. The heparanase enzyme is a promising target for development of new anticancer drugs. HS and the structurally related heparin are present in most animal species. As an analogue of the natural substrate of heparanase HS, heparin is considered to be a potent inhibitor of heparanase. SST0001 is a polymer with a heparin-like structure. It is a reduced oxidized N-acetyl heparin, these modifications cause the reduction of anticoagulant activity and are strictly related to the anti-heparanase activity. In preclinical murine models SST0001 showed a significant anti myeloma effect in multiple myeloma mice xenograft models, with a significant reduction of subcutaneous growth of different multiple myeloma cell lines, when SST0001 was administered either alone or in combination with dexamethasone. The purpose of this study is to determine the safety and tolerability of escalating doses of SST0001 in the treatment of advanced refractory multiple myeloma.

DETAILED DESCRIPTION:
Multicenter, open label, uncontrolled Phase I First In Man trial in advanced refractory multiple myeloma, to determine the Maximum Tolerated Dose (MTD) of SST0001 given subcutaneously (sc) once daily for 5 or 10 days, in a cycle of 28 days. A starting dose of 25 mg (flat dose) is given once daily for 5 days (from Day 1 to Day 5). In the subsequent cohort 25 mg are administered once daily for 10 days (from Day 1 to 5 and from Day 8 to 12). Dose escalation with SST0001 administered for 10 days is performed in subsequent cohorts, depending on toxicities observed.

Indirect pharmacokinetics based on Activated Partial Thromboplastin Time (aPTT) modifications in all patients (minimum of 3 patients in each cohort) during the first cycle of treatment and direct SST0001 concentrations measurements.

Pharmacodynamics in all patients during the first cycle of treatment, based on modifications of coagulation parameters.

During the study any hints of anti-tumor activity will also be evaluated based on use of surrogate parameters (monoclonal serum and urine protein modifications).

ELIGIBILITY:
Inclusion Criteria:

* Advanced, heavily pretreated refractory multiple myeloma (MM).
* Patient should have exhausted all available anti MM therapies.
* Age ≥18 years.
* ECOG (Eastern Cooperative Oncology Group)performance status ≤ 2.
* Life expectancy of more than 3 months.
* No concomitant use of anticoagulants or antiplatelets drugs such as aspirin, NSAIDs (Nonsteroidal Antiinflammatory Drug), Clopidogrel, Unfractionated Heparin, Low Molecular Weight Heparin (e.g. Enoxaparin), Fondaparinux, Dabigatran, Rivaroxaban, Apixaban and Warfarin.
* No platelets diseases or allergy to anticoagulants.
* WBC (White Blood Cell) ≥2000/µL; Platelets ≥50,000/µL; Hb ≥ 8 g/dL.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST (aspartate aminotransferase)and ALT (alanine aminotransferase)≤ 3 x the ULN; serum creatinine ≤ 1.5 x the ULN (Upper Limit of Normal).
* aPTT, TT, INR, fibrinogen, D-dimer within ULN.
* Disease free of prior malignancies for ≥ 3 years.
* No acute gastrointestinal bleeding or any major bleeding (e.g CNS) in the past 2 years or any significant bleeding history.
* No known central nervous system involvement by myeloma.
* Capacity of understanding the nature of the trial and giving written informed consent.
* Unless a female patient is post-menopausal or surgically sterilized, must be willing to use an acceptable method of birth control (hormonal contraceptive, intrauterine device, barrier contraceptive with spermicide, or abstinence) for the duration of the study.
* Male patient must agree to use an acceptable method for contraception (barrier contraceptive or abstinence) for the duration of the study.

Exclusion Criteria:

* Pregnancy or lactation or unwillingness to use adequate method of birth control
* Ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients.
* Active uncontrolled viral, bacterial, or fungal infection or history of HIV, hepatitis B or C, or any infection requiring systemic antivirals or antimicrobials.
* Grade ≥ 2 toxicity due to previous anti-neoplastic therapy (except alopecia), and Grade ≥ 3 peripheral motor or sensory neuropathy, in the 2 weeks before treatment (CTCAE V4.0).
* Less than 2 weeks since most recent chemotherapy, or concurrent chemotherapy.
* Presence of cirrhosis or chronic hepatitis.
* Diagnosis of amyloidosis or diagnosis of plasma cell leukaemia.
* Presence of serious cardiac (congestive heart failure, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorder.
* Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD). | 28 days of first cycle of therapy.
  Maximum tolerated dose (MTD) (based upon first cycle study drug related dose limiting toxicities [DLTs]) of SST0001 given subcutaneously over repeated administration during each treatment cycle. MTD definition: ≥ 2/6 patients with a DLT at the first cycle (28 days).

SECONDARY OUTCOMES:
Adverse events, physical examination and laboratory tests. | 28 days of each cycle of therapy.
  Number of patients with adverse events, number of patients with abnormalities at physical examination and laboratory tests (hematology and biochemistry) as a measure of safety and local tolerability of SST0001. Safety assessments and severity of adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) V4.0.
Maximum plasma concentration (Cmax) | 28 days of first cycle of therapy.
  Blood pharmacokinetics of SST0001 using Activated Partial Thromboplastin Time (aPTT)as indirect measurement of SST0001 equivalent plasma concentrations.
Time to achieve Cmax (Tmax) | 28 days of first cycle of therapy.
Area under the concentration curve from administration to the last observed concentration time (AUClast) | 28 days of first cycle of therapy.
Half-life (T1/2) | 28 days of first cycle of therapy.
aPTT (Activated Partial Thromboplastin Time) | 28 days of first cycle of therapy.
  Pharmacodynamics of SST0001 in terms of effects on coagulation profile (aPTT, seconds).
TT (Thrombin Time) | 28 days of first cycle of therapy.
  Pharmacodynamics of SST0001 in terms of effects on coagulation profile (TT, seconds).
INR (International Normalized Ratio) | 28 days of first cycle of therapy.
  Pharmacodynamics of SST0001 in terms of effects on coagulation profile (INR).
Tumor response. | 28 days of each cycle of therapy.
  Antitumor activity through the use of surrogate parameters (monoclonal serum and urine protein modifications), by means of serum and urine protein electrophoresis, immunoelectrophoresis and immunofixation, Serum Free Light Chain (FLC) Ratio and/or 24-h Bence-Jones urine protein.
  M-protein (g/dL), Bence-Jones protein (g/24h), kappa FLC (mg/dL) and lambda FLC (mg/dL) will be assessed at each cycle of therapy. Responses will be evaluated according to International Myeloma Working Group (IMWG) Guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — USC Ematologia, Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Italy; Arnon Nagler, MD, Principal Investigator — Division of Hematology, Chaim Sheba Medical Center, Tel Hashomer, Israel; Manik Chatterjee, MD, Principal Investigator — Universitätsklinik Würzburg, Medizinische Klinik und Poliklinik II (ZIM), Würzburg, Germany
Locations (5):
- Manik Chatterjee, Würzburg, Germany
- Division of Hematology, Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (3):
  - U.O. Ematologia con Trapianto, Dipartimento dell'Emergenza e dei Trapianti di Organi, Bari
  - USC Ematologia, Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - S.C. Ematologia, ASO S. Croce e Carle - Cuneo, Cuneo